CLINICAL TRIAL: NCT01953393
Title: The Acute Effects of Low-dose TNF-α on Glucose Metabolism and β-cell Function in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Tobias Ibfelt, MD, Rigshospitalet, Denmark
Purpose: Basic Science
Other Study IDs: RH TAL
Record Dates: First submitted 2013-09-13; First posted 2013-10-01 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-09

CONDITIONS: Diabetes Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Tumor Necrosis Factor-alpha

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Low-dose TNF-alpha

SUMMARY:
Type 2 diabetes is characterized by increased insulin resistance and impaired insulin secretion. In addition, type 2 diabetes is associated with low grade inflammation indicated by increased levels of proinflammatory cytokines such as TNF-α. TNF-α has previously been shown to impair peripheral insulin signaling in vitro and in vivo. However, it is unclear whether TNF-α may also affect endogenous glucose production (EGP) during fasting and glucose stimulated insulin secretion (GSIS) in vivo.

We hypothesized that low dose TNF-α would increase EGP and attenuate GSIS. Recombinant human TNF-α or placebo was infused in healthy, non-obese and non-diabetic young men (n=10) during a 4-hour basal period followed by an intravenous glucose tolerance test (IVGTT).

ELIGIBILITY:
Inclusion Criteria:

* Healthy men
* Age 20-35

Exclusion Criteria:

* obesity (BMI>25)
* diabetes
* chronic disease

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2006-04; Primary Completion 2006-05 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Beta-cell function | Measurements at 0h, 1h, 2h, 3h and 4h during basal period. After glucose bolus infusion, measurements every 1 min for the first 30 min and every 3 mins for the next hour. Last measurement 1,5 hours post- IVGTT
  Insulin levels (pg/ml) in blood measured continually before and after Intravenous glucose tolerance test. Glucose bolus infused in healthy young men after a 4 hour basal period. Subsequent measurements og insulin and glucose levels in peripheral blood

CONTACTS AND LOCATIONS:
Overall Officials: Christian P Fischer, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- 1 The Centre of Inflammation and Metabolism, Department of Infectious Diseases and CMRC, Rigshospitalet, Faculty of Health Sciences, University of Copenhagen, Copenhagen N, Denmark

REFERENCES:
- [Result] Plomgaard P, Fischer CP, Ibfelt T, Pedersen BK, van Hall G. Tumor necrosis factor-alpha modulates human in vivo lipolysis. J Clin Endocrinol Metab. 2008 Feb;93(2):543-9. doi: 10.1210/jc.2007-1761. Epub 2007 Nov 20. PMID 18029463